CLINICAL TRIAL: NCT06948123
Title: The Effect of Nursing Approach Based on MELEIS Transition Theory on Cardiac Quality of Life and Adaptation to Disease in Patients With Acute Myocardial Infarction
Brief Title: Myocardial Infarction
Acronym: Nursing Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Serdar Zengin, internal medicine nursing PhD, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMU-HEM-SZ-01
Record Dates: First submitted 2025-03-17; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndromes
Keywords: acute coronary syndrome; transition theory; Nursing Caries
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Early Intervention, Educational; Control Groups

STUDY DESIGN:
Intervention Model Description: This research was conducted with two groups as experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-based nursing intervention. (Experimental): This is the group that was trained with educational material prepared by the researcher based on Meleis's Transition Theory.
  Interventions: Other: Educational intervention
- Control (Other): The control group was visited at home 15 days after discharge and the scales were applied. The final scales were applied to the patient who came to the hospital for 3 months. The patient was told that the study was over and given educational materials.
  Interventions: Other: control group

INTERVENTIONS:
Other: Educational intervention — The experimental group was trained with educational material prepared by the researcher using a computer at home for 15 days after hospital discharge.
  Arms: Theory-based nursing intervention.
Other: control group — The control group was visited at home 15 days after discharge and the scales were applied. The final scales were applied to the patient who came to the hospital for 3 months. The patient was told that the study was over and given educational materials.
  Arms: Control

SUMMARY:
The effect of nursing approach based on Meleis's transition theory on cardiac quality of life and adaptation to disease in patients with acute myocardial infarction.

This research was planned with the idea that the approach developed based on Meleis's Transition Theory could facilitate the illness-health transition process in patients, increase their healthy behavioral gains, increase the quality of care, reduce rehospitalizations, reduce the mortality rate due to MI, and contribute to the nursing literature.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is one of the important health problems with high morbidity and mortality in the world and in our country. More than 9 million people die due to CAD every year in the world, and this condition constitutes 14.8% of all deaths . TEKHARF study data in 2017 show that CAD mortality and prevalence are higher in Turkish adults compared to European countries. Myocardial infarction (MI) is defined as CAD that develops due to prolonged ischemia and shows clinical features including electrocardiographic findings, elevation of biochemical markers of myocardial necrosis, and imaging. According to 2015 data of the American Heart Association, the prevalence of MI is 3.3% in men and 1.8% in women aged 40-59; It was announced as 11.3% in men and 4.2% in women between the ages of 60-79. When looking at the 2018 data of the Turkish Statistical Institute (TUIK), circulatory system diseases are in the first place with 38.4% (162 thousand) of all death cases (423 thousand). Ischemic heart disease constitutes 39.7% of deaths due to circulatory system diseases . In the Heart Disease Risk Factors in Turkish Adults study, the annual CAD death rate in European countries was reported as 2 to 8 per thousand in men and 0.6 to 3 per thousand in women between the ages of 45-74. In our country, this rate was found to be 7.6 per thousand in men and 3.8 per thousand in women in the same age range . According to the data of the Ministry of Health, the incidence of myocardial infarction is stated as 156,300 per hundred thousand and its prevalence as 0.648 per thousand. MI is generally seen as an important health problem that is difficult to adapt to because it is more common in the productive age group, causes serious problems such as post-acute rhythm problems, development of heart failure, recurrence of MI, ischemia, ventricular fibrillation, post-infarction angina, causes loss of work force, and has a negative impact on quality of life and the economic burden it brings. Social, psychological and physical limitations after MI negatively affect individuals' quality of life and self-efficacy levels and make compliance difficult . Studies have shown that patients have difficulty in making lifestyle changes after MI, and this increases the risk of re-infarction . The study conducted by Ens and colleagues (2019) also states that most patients who have had MI do not know cardiovascular disease risk factors, symptoms and how to make lifestyle changes. In another study on compliance with medication use, it was found that a significant portion of patients with acute coronary syndrome after MI had impaired treatment compliance after one year. The main goal in the treatment of MI is to prevent cardiac recurrence and complications and to adapt to lifestyle changes. Lifestyle changes in the management of myocardial infarction risk factors (smoking, alcohol, obesity, hyperlipidemia, hypertension, diabetes, physical activity, weight control and diet) are emphasized by the American Heart Association and the European Society of Cardiology. Lifestyle changes after MI reduce the risk of infarction and mortality. International guidelines emphasize that exercise programs after myocardial infarction reduce the mortality rate by 20%, smoking cessation reduces the risk of a new infarction by 50%, and dietary changes and the use of lipid-lowering drugs reduce the risk of a new infarction by 34% and total mortality by 30%. . It is reported that ensuring compliance will be important for patients to return to their active lives and continue their lives in a healthy way after MI. Many interventions such as home visits, telephone follow-up and motivational interviews, increasing self-management, providing education and counseling are used to increase compliance and quality of life. Among these interventions, education is reported to be an effective method in increasing awareness and responsibility, contributing to lifestyle changes, and telephone follow-up is an effective method in increasing quality of life and self-efficacy, reducing stress, and preventing repeated hospitalizations . It is stated that theory-based interventions are effective in increasing the effectiveness of nursing interventions . One of these theories is the theory of transitions founded by Meleis. Meleis defines transitions as new situations that occur as a result of changes in life, health, illness, personal and social relationships . Being diagnosed with a disease, becoming a mother, taking on a new task, changing profession, being hospitalized or discharged are all situations that involve transitions. Change and development are extremely important for nursing, and transitions are always related to these two concepts . Nursing often involves clients and their families in various types of transitions and determines the changes that transitions create in the lives of clients and their families and the nursing care needs, and plans and implements the necessary interventions. Therefore, transition theory generally emerges as a theory that systematically and comprehensively displays nursing phenomena related to transitions . When transitions are related to health or illness or when the responses to the transition are related to health-related behaviors, these transitions fall within the scope of nursing . Nurses tend to be caregivers who prepare their clients for upcoming transitions and teach them coping mechanisms that facilitate the process of learning new skills related to their health and illness experiences. In transition theory, four types of transitions have been defined, based on the experiences of nurses working with patients and their families: developmental, situational, health-illness, and institutional. Health-disease transitions include sudden changes that cause sudden or gradual transitions from a state of wellness to a state of illness, or from a state of illness to a state of health . Early assessment of process indicators in transitions that facilitate health or increase vulnerability is necessary for the development of interventions that facilitate healthy outcomes . In a study conducted in our country on individuals newly diagnosed with diabetes using the transition theory, it was determined that there was a significant increase in patients' self-management and adaptation to the disease . In another study conducted based on the transition theory to increase the quality of life in menopause, it was determined that the quality of life increased . In another study using the transition theory, it was determined that the quality of care during discharge increased, and health care costs decreased with fewer readmissions. In another study conducted on elderly individuals with cognitive impairment, it was determined that the cost of the Transition Care Model was low . No randomized controlled study has been found in the literature using education and digital monitoring based on Meleis's transition theory in improving the quality of life and compliance with lifestyle changes in patients who have had an MI. This research was planned with the idea that the approach developed based on Meleis's Transition Theory could facilitate the illness-health transition process in patients, increase their healthy behavioral gains, increase the quality of care, reduce rehospitalizations, reduce the mortality rate due to MI, and contribute to the nursing literature.

ELIGIBILITY:
Inclusion Criteria:

Among the patients who were hospitalized in the Cardiology Clinic of Aydın State Hospital and underwent emergency coronary angiography;

* Those who were 18 years of age and older, diagnosed with MI,
* Underwent coronary angiography for the first time,
* Conscious,
* No verbal communication barrier,
* Able to read and write,
* Had their polyclinic check-ups at the relevant hospital,
* Agreed to participate in the study,
* Had a telephone to communicate,
* Living in Aydın city center and districts were included in the study.

Exclusion Criteria:

* Patients with COPD,
* Chronic renal failure,
* Cancer, arrhythmia,
* Advanced aortic stenosis and pulmonary hypertension,
* Systemic or pulmonary embolism,
* Chronic cognitive and psychiatric diseases,
* Patients scheduled for organ transplantation,
* Ptage 3 and 4 heart failure (according to New York Heart Association standards),
* Patients with a hospital stay longer than 10 days were excluded from the study

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Psychosocial Adjustment-Self-Report Measure (PAIS-SR ), | 3 months for each patient.
  Psychosocial Adjustment-Self-Report Measure: PAIS-SR: This scale assesses psychological adjustment to illness. Cronbach's alpha coefficient for the overall scale has been reported to be 0.92. The scale consists of 46 items and seven subscales. A total score of less than 35 indicates "good psychosocial adjustment," a score between 35 and 51 indicates "moderate psychosocial adjustment," and a score greater than 51 indicates "poor psychosocial adjustment."
Health-related Quality of Life scale (HEART-QOL) | 3 months for each patient.
  HEART-QOL: A tool developed to measure quality of life specific to heart disease. The questionnaire is a scale consisting of 27 items and 7-point Likert type responses, and has 3 sub-dimensions: emotional, physical and social. Scores are calculated by taking the average of the items for each dimension. Scores range from 1 to 7, with a low score indicating poor quality of life and a high score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: RAHŞAN ÇEVİK AKYIL, PROFESSOR, Study Director — Aydin Adnan Menderes University Faculty of Nursing
Locations (1):
- Aydin State Hospital, Aydin, AYDIN/Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to disclose the work as I will publish it myself at certain times.